CLINICAL TRIAL: NCT05667168
Title: Physiotherapeutic Diagnostic and Therapy of Tinnitus
Brief Title: Physiotherapeutic Approach to Tinnitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Charles University, Czech Republic (Other)
Collaborators: The Jerzy Kukuczka Academy of Physical Education in Katowice (Other)
Responsible Party: Principal Investigator, Malá Jitka, Clincial Professor, Charles University, Czech Republic
Allocation: Non-Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: FTVS
Record Dates: First submitted 2022-12-19; First posted 2022-12-28 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2022-12

CONDITIONS: Tinnitus
Keywords: headache; noise; laser; manual therapy; temporomandibular dysfunction
MeSH Terms: conditions — Tinnitus; Headache; Temporomandibular Joint Disorders

STUDY DESIGN:
Intervention Model Description: intervention study
Who Masked: Participant, Care Provider
Masking Description: The participants and care providers will not know the checking data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- High power laser (Experimental): The application of high-intensity laser on cervical muscles, 50J/cm2, 980nm, 0 Hz, on processus mastoideus and porus acusticus externus.
  Administration of tinnitus intensity on scale 0-10 and questionary.
  Interventions: Procedure: physiotherapy approach
- Low power laser (Experimental): The application of low-intensity laser on cervical muscles, 4J/cm2, 980nm, 0 Hz, on processus mastoideus and porus acusticus externus. Administration of tinnitus intensity on scale 0-10 and questionary.
  Interventions: Procedure: physiotherapy approach
- Radio-frequention therapy (Experimental): Applying radio-frequentation current on cervical muscles, 10-50% of intensity, 0 Hz. Administration of tinnitus intensity on a scale of 0-10 and questionary.
  Interventions: Procedure: physiotherapy approach
- Manual therapy of temporomandibular joint,. (Experimental): A manual physiotherapeutic approach to the temporomandibular joint will treat participants. Administration of tinnitus intensity on a scale of 0-10 and questionary.
  Interventions: Procedure: physiotherapy approach
- Manual therapy of the cervical spine. (Experimental): A manual physiotherapeutic approach to the cervical spine will treat participants. Administration of tinnitus intensity on a scale of 0-10 and questionary.
  Interventions: Procedure: physiotherapy approach
- Physical exercising. (Active Comparator): Participants will be treated by physical exercising in closing and opening muscle chains. Administration of tinnitus intensity on a scale of 0-10 and questionary.
  Interventions: Procedure: physiotherapy approach
- Cognitive therapy (Active Comparator): Participants will be treated with cognitive therapy by a psychologist. Administration of tinnitus intensity on a scale of 0-10 and questionary.
  Interventions: Procedure: physiotherapy approach
- Life style. (Placebo Comparator): Participants will be treated only by modulation of their lifestyle. Administration of tinnitus intensity on a scale of 0-10 and questionary.
  Interventions: Procedure: physiotherapy approach

INTERVENTIONS:
Procedure: physiotherapy approach — The therapy will take place 2-3 times a week; the therapeutic unit will last 45 minutes and will be oriented towards one therapeutic approach from the above list. The total number of therapy sessions will be limited to 3 months (i.e. three months, 2-3 times a week). After completion of the 3-month therapy, a follow-up examination will be performed again by kinesiological analysis, questions about the intensity of tinnitus according to a numerical scale and quality of life by a selected questionnaire.

SUMMARY:
Intervention experiments in the physiotherapeutic field targeted diagnostics and therapy of tinnitus. The goal is to find various groups of tinnitus patients and an ideal therapeutic approach between physical therapy means, manual techniques and physical education approach.

DETAILED DESCRIPTION:
Clients will be divided into individual (8) therapy groups. The proband groups formed will be treated by individual researchers according to a similar methodology, each with a different therapeutic intervention for tinnitus. The main dominant variables to be monitored will be tinnitus intensity assessed on a visual numerical scale from 0-10, and quality of life observed using different questionnaires (which questionnaires will be used will be addressed in the course of the research, as this is not standardly used for tinnitus in the Czech region). The questionnaires will measure the quality of life and intensity of tinnitus of probands at the beginning and the end of the experiment, regardless of their racial, political, social, religious, and philosophical views and classification. Sexual orientation and criminal offences will not be questioned or addressed. As part of the questionnaires, clients will be subjected to musculoskeletal diagnosis by kinesiological analysis and tinnitus diagnosis by examination and will be further assigned to appropriate therapy sections (8). The questionnaires will be given to probands in hard copy at the initial assessment, during which the proband will complete and submit the questionnaire. The exit questionnaire will be administered similarly at the exit examination, i.e. the proband's last visit to the research team.

The selected therapeutic interventions in each section will be a low-power laser, high-power laser, radiofrequency therapy, manual therapy of the temporomandibular joint, manual treatment of the cervical and adjacent thoracic spine, myofascial chain work in the context of closed and open kinematic patterns, psychological guidance mediated by a psychosomatic physician, and addressing healthy lifestyle issues. The therapy will take place 2-3 times a week; the therapeutic unit will be 45 min and will be oriented to one therapeutic approach from the above list. The total number of therapy sessions will be limited to 3 months (i.e. three months, 2-3 times a week). The therapy will take place at the clinical workplace of private practice (anonymise) and the practice rooms of the Department of Physiotherapy Faculty of Physiotherapy of Charles University. At the end of the 3-month therapy, a follow-up examination will be performed again by kinesiological analysis, questions about the intensity of tinnitus according to a numerical scale and quality of life by a selected questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* neurologically diagnosed tinnitus
* age 20-80 years
* tinnitus of any nature persisting for more than 3 months

Exclusion Criteria:

* acute or chronic medical conditions requiring medication
* history of head and cervical spine trauma
* oncologic therapy
* psychological or psychiatric treatment

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-25 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Decreasing of sensoric feeling of tinnitus. | 3 month
  Due to analog numeric scale (0-10 where 0 mean without tinnitus and 10 maximum intensity of tinnitus), will be find the most effective approach to decreasing hearable sound typical for tinnitus.
Changing of life quality due to tinnitus. | 3 month
  According to the questionnaire survey (THI) the effect of the treatment will be shown.

CONTACTS AND LOCATIONS:
Overall Officials: Jitka Malá, PhD., Study Director — Charles University Prague, Czech Republic
Locations (1):
- Charles University, Faculty of physical education and sport, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No